CLINICAL TRIAL: NCT04633902
Title: Phase II Study of Olaparib in Combination With Pembrolizumab in Patients With Advanced Melanoma With Homologous Recombination (HR) Pathway Gene Mutation
Brief Title: Phase II Study of Olaparib and Pembrolizumab in Advanced Melanoma With Homologous Recombination (HR) Mutation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: California Pacific Medical Center Research Institute (Other)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPMC19-MEL01
Record Dates: First submitted 2020-11-12; First posted 2020-11-18 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Metastatic Melanoma
Keywords: Homologous recombination (HR); Mutation; Olaparib; Pembrolizumab; PARP inhibitor; anti PD-1 antibody
MeSH Terms: conditions — Melanoma | interventions — olaparib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Olaparib + Pembrolizumab (Experimental): This arm will enroll patients who has advanced melanoma with a genetic HR mutation/ alteration including mutation/ deletion in ARID1A/B, ARID2, ATM, ATR, BARD1, BRCA1/2, BAP1, BRIP1, CHEK2, FANCA, FANCD2, MRN11A, PALB2, RAD50, RAD51, RAD54B.
  Interventions: Drug: Olaparib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Olaparib — Olaparib 300 mg BID daily
  Other Names: Lynparza
Drug: Pembrolizumab — Pembrolizumab 200 mg IV eveyr 3 weeks (for up to 2 years)
  Other Names: Keytruda

SUMMARY:
This open-label phase II trial studies how well olaparib in combination with pembrolizumab works in treating patients with advanced, metastatic melanoma with the homologous recombination (HR) pathway gene mutation / alteration. Olaparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth, and potentially augment an anti-tumor immune response to pembrolizumab. The trial is designed to assess the efficacy and safety of olaparib in combination with pembrolizumab in patients with HR mutation/ alteration whose disease progressed on prior immunotherapy and/or BRAF-targeting therapy

DETAILED DESCRIPTION:
Treatment with PARP inhibitors could represent a novel opportunity to selectively kill a subset of cancer cells with deficiencies in DNA repair pathways. For example, a tumor arising in a patient with a germline BRCA mutation (gBRCAmut) has a defective homologous recombination DNA repair pathway and would be increasingly dependent on NHEJ, alt-NHEJ, and BER for maintenance of genomic integrity. PARP inhibitors block alt-NHEJ and BER, forcing tumors with BRCA deficiencies to use the error-prone NHEJ to fix double-strand breaks. Non-BRCA deficiencies in homologous recombination DNA repair genes could also enhance tumor cell sensitivity to PARP inhibitors. The rationale for anticancer activity in a subset of non-gBRCAmut tumors is that they share distinctive DNA repair defects with gBRCAmut carriers, a phenomenon broadly described as "BRCAness." DNA repair defects can be caused by germline or somatic alterations to the homologous recombination DNA repair pathway. Homologous recombination is a complex pathway, and several genes other than BRCA1 and BRCA2 are required either to sense or repair DNA double-strand breaks via the homologous recombination pathway. Therefore, PARP inhibitors are also selectively cytotoxic for cancer cells with deficiencies in DNA repair proteins other than BRCA1 and BRCA2.

In melanoma, genetic HR mutation/ alterations are rather common. Retrospective data showed that nearly 20-30% of cutaneous melanoma harbors a mutation in at least 1 of the HR genes in their tumor. The commonly altered genes were ARID1A, FANCA, ATM, BRCA1, ATRX and BRCA2, ATR, BRCA1 and BRIP1. These findings indicate that HR mutations / alterations are frequently observed in metastatic melanoma, and they suggest that PARP inhibitors could potentially be of a great clinical value in a substantial portion of the patients with advanced melanoma. In addition, the retrospective data also showed that presence of HR mutation was associated with high TMB and clinical response to checkpoint immunotherapy. Therefore, the investigators propose a phase II study of niraparib in patients with advanced melanoma with genetic homologous recombination mutation/ alteration.

In this clinical study, clinical efficacy of olaparib in combination with pembrolizumab will be evaluated by assessing an objective clinical response rate in patients with advanced, metastatic melanoma with the homologous recombination (HR) pathway gene mutation / alteration. All participating patients will receive olaparib 300 mg a day and pembrolizumab 200 mg every 3 weeks (for up to 2 years) until disease progresses or they experience intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of unresectable or metastatic stage III or IV melanoma
* Must have genetic HR mutation/ alteration including ARID1A/B, ARID2, ATM, ATR, BARD1, BRCA1/2, BAP1, BRIP1, CHEK2, FANCA, FANCD2, MRN11A, PALB2, RAD50, RAD51, RAD54B
* Disease must be refractory or resistant to anti PD-1 therapy (defined as disease progression within 6 months after the last dose of anti PD-1 antibody therapy) and, for V600 BRAF mutation, disease must be progressed after BRAF inhibitor therapy; or patients could not have tolerated the standard therapies.
* Must have measurable disease based on RECIST 1.1.
* Must have an ECOG performance status of 0 to 1.
* Prior systemic cytotoxic therapy up to 1 regimens is allowed; There is no limit on the number of prior immunotherapy or targeted therapy regimens.
* Must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline.

Exclusion Criteria:

* Previously treated with a PARP inhibitor
* Has received prior radiotherapy within 2 weeks of start of study treatment. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has a known additional malignancy that is progressing or has required active treatment within the past 2 years
* Previous solid organ or allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT) for solid tumors.
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
* Has active autoimmune disease that has required systemic treatment in the past 2 years
* Has a history of (non-infectious) pneumonitis due to a single agent PD-1 / PD-L1 antibody therapy that required steroids or has current pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 6 months
  ORR of olaparib in combination with pembrolizumab in patients with advanced melanoma with genetic homologous recombination (HR) mutation/ alteration using RECIST v1.1

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 2 years
  PFS of patients with advanced melanoma with genetic HR mutation/ alteration who are treated with olaparib in combination with pembrolizumab
Overall survival (OS) | 2 years
  OS of patients with advanced melanoma with genetic HR mutation/ alteration who are treated with olaparib in combination with pembrolizumab
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | 2 years
  Evaluation of the safety profile of olaparib in combination with pembrolizumab in patients with advanced melanoma with genetic homologous recombination (HR) mutation/ alteration

CONTACTS AND LOCATIONS:
Overall Officials: Kevin B Kim, MD, Principal Investigator — California Pacific Medical Center Research Institute
Locations (2):
- United States (2):
  - California Pacific Medical Center Research Institute, San Francisco, California
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No